CLINICAL TRIAL: NCT00790829
Title: Preemptive Use of Nicotine Patch for Postoperative Pain Relief in Open Abdominal Surgery
Brief Title: Preemptive Use of the Nicotine Patch for Postoperative Pain Relief After Open Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Ursula Landman, principal investigator, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20075594
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2011-08

CONDITIONS: Postoperative Pain
Keywords: preemptive; Nicotine Patch; Open Abdominal Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Tobacco Use Cessation Devices; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A, B (Experimental): Group B received a seven-milligram transdermal patch and Group A received a placebo patch.
  Interventions: Drug: transdermal nicotine patch

INTERVENTIONS:
Drug: transdermal nicotine patch — Generic seven-milligram nicotine patches for 24hours, placebo patch for 24 hours
  Other Names: Generic

SUMMARY:
The efficacy of a low dose nicotine patch of seven milligrams placed before surgery and its effect on decreasing pain after surgery is the main purpose of the study.

DETAILED DESCRIPTION:
Study patients include nonsmokers aged 18-75 undergoing open abdominal wall surgery under general anesthesia. If the patient smokes, receives a regional anesthetic such as an epidural, or is pregnant, then he/she is excluded from the study. There are two randomized study groups. Group B receives a seven-milligram transdermal patch and Group A receives a placebo patch. Generic seven-milligram nicotine patches or identical placebo patches made from band-aids are glued to a 3x4 inch adhesive pad and placed on the individuals' right upper arm 1 hour before surgery. All patients are given a standardized anesthetic consisting of a narcotic infusion, propofol, a neuromuscular blocking agent, anesthetic gas agent, antinauseant medication and a nonsteroidal.

Patients receive postoperative analgesia for twenty four hours after surgery with a narcotic or an additional nonsteroidal medication. All patients receive intravenous controlled patient controlled analgesia (IVPCA) with morphine sulfate one milligram per ten minutes, forty milligram four hour limit. Patients also receive toradol fifteen milligrams for breakthrough pain. The patch is removed from participants twenty four hours post IVPCA initiation. The following items are assessed every four hours for twenty four hours after post anesthesia care unit discharge: a verbal rating of pain, total IVPCA morphine use, nausea occurrence, vomiting occurrence, and sedation score by the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Study patients include nonsmokers aged 18-75 undergoing open abdominal wall surgery under general anesthesia.

Exclusion Criteria:

* If the patient smokes, receives a regional anesthetic such as an epidural, or is pregnant, then he/she is excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of a low dose nicotine patch of seven milligrams placed before surgery and its effect on decreasing pain after surgery is the main purpose of the study. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ursula N Landman, DO, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States